CLINICAL TRIAL: NCT01675609
Title: A Single-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of Brimonidine Tartrate Ophthalmic Solution in Adult and Geriatric Subjects
Brief Title: Study Evaluating the Safety and Efficacy of Brimonidine Tartrate Ophthalmic Solution in Adult and Geriatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eye Therapies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-100-0015
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Ocular Redness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Brimonidine Tartrate 0.025% (Experimental)
  Interventions: Drug: Brimonidine tartrate 0.025%

INTERVENTIONS:
Drug: Placebo — 1 drop in each eye daily for up to 35 days
  Arms: Placebo
Drug: Brimonidine tartrate 0.025% — 1 drop in each eye for up to 35 days
  Arms: Brimonidine Tartrate 0.025%

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of brimonidine tartrate 0.025% ophthalmic solution used four times daily in a population of adult and geriatric subjects

ELIGIBILITY:
Inclusion Criteria:

* Be at least 40 years of age
* Must have normal ocular health
* Must have history of redness relief drop use or desire to use

Exclusion Criteria:

* Must not have any ocular/systemic health problems
* Must agree to avoid disallowed medications

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Ocular redness | at specified timepoints for up to 180 minutes
  redness evaluated by investigator prior to study medication instillation and redness evaluated by the subject as captured in dosing diary

SECONDARY OUTCOMES:
Ocular Redness | up to 5 minutes post study medication instillation
  evaluated prior to study medication instillation and at 5 minutes post instillation

CONTACTS AND LOCATIONS:
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States